CLINICAL TRIAL: NCT03198897
Title: BioHoFH - Biomarker for Homozygous Familial Hypercholesterolemia AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Homozygous Familial Hypercholesterolemia (BioHoFH)
Acronym: BioHoFH
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BHFH 06-2018
Record Dates: First submitted 2017-06-19; First posted 2017-06-26 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Lipoprotein Lipase Deficiency; Inborn Error of Lipid Metabolism; Corneal Arcus
Keywords: familial hypercholesterolaemia; Biomarker
MeSH Terms: conditions — Hyperlipoproteinemia Type I; Lipid Metabolism, Inborn Errors; Arcus Senilis; Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectrometry, a blood sample will be taken vis using a dry blood spot filter card and will be analysed in a specialist laboratory. To proof the correct diagnosis a homozygous familial hypercholes-terolemia, in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of a homozygous familial hypercholesterolemia will be per-formed. The analyses will be done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with a Homozygous familial Hypercholesterolemia or high-grade suspicion for Homozygous familial Hypercholesterolemia

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Homozygous familial Hypercholesterolemia from blood

DETAILED DESCRIPTION:
Homozygous familial hypercholesterolemia (HoFH) is a rare hereditary disorder of lipoprotein metabolism characterized by exceptionally high levels of low-density lipoprotein cholesterol (LDL-C). Clinical manifestations may vary but often include markedly premature coronary artery disease, supravalvular aortic stenosis due to aortic root atheroma, and cutaneous manifestations such as tendon xanthomata. Although there are no universally ac-cepted clinical diagnostic criteria for HoFH, an untreated serum LDL-C of >13 mmol/L (500 mg/dL), or an on-treatment LDL-C of more 8 mmol/L (300 mg/dL) together with the appearance of cutaneous xanthomata before the age of 10 years, have often been used to diagnose HoFH clinically. As molecular diagnostic techniques have advanced, genotyping of patients with severe hypercholesterolemia has become an integral part of clinical practice in many settings. This has led to the realization that the spectrum of clinical severity in HoFH is much wider than initially thought and that the clinical criteria often fail to identify patients with milder phenotypes.

Although the HoFH phenotype may result from mutations in multiple genes, low-density lipoprotein receptor (LDL-R) dysfunction is the final common pathophysiological pathway leading to LDL-C elevation in patients with HoFH and LDL-R mutations are by far the most common genetic causes of HoFH. Patients with HoFH secondary to LDL-R mutations inherit a mutated allele from each parent, resulting in severe functional impairment of the LDL-R pathway. Residual LDL-R activity may vary considerably between mutations. Patients with HoFH can be classified as receptor negative or receptor defective (<2% or 2%-25% of residual activity, respectively) based on LDL uptake studies in cultured fibroblasts, although receptor function is nowadays often inferred after the identification of specific mutations.

Historically, the prevalence of HoFH has been reported as 1 case per million. However, emerging studies suggest that the prevalence of HeFH, and consequently HoFH, may be higher than previously thought. Recent literature suggests an estimated prevalence of HeFH of ∼1 case in 2002 and of deleterious LDLR mutations in 0.45% of a control population and 1.9% of individuals with early-onset myocardial infarction or coronary artery dis-ease.Extrapolating from these data, the prevalence of HoFH is estimated to be ∼6 cases per million. Analysis of a Dutch database of molecularly defined HoFH suggested a prevalence of ∼1 case per 160,000-300,000. Prevalence data are, however, continuing to evolve, and these calculations could be underestimates or overestimates of the prevalence in the general patient population. Information on the prevalence of FH in non-European populations is generally limited, and conclusions about the possible worldwide prevalence remain speculative. However, as a result of founder effects, the prevalence of HeFH and HoFH is higher in certain populations such as the Afrikaners in South Africa, Christian Lebanese, and French Canadians.

The range of untreated and treated LDL-C levels in HoFH is wide. In two recent clinical tri-als of novel therapies for HoFH, the LDL-C levels at study entry in conventionally treated patients ranged from a mean of 8.7 ± 2.9 mmol/L (336 ± 112 mg/dL) to 11.4 ± 3.6 mmol/L (441 ± 139 mg/dL). Not all patients with HoFH have extreme LDL-C elevations. In a study from the Netherlands, only 50% of patients with molecularly defined HoFH met the clinical criterion of untreated LDL-C >13 mmol/L (500 mg/dL), with some patients presenting with untreated LDL-C levels as low as 4.4 mmol/L (170 mg/dL).

Reported LDL-C levels for clinical and genetic diagnoses of FH. Improved molecular diagnosis has led to the understanding that a conventional diagnosis of HoFH encompasses a wide range of underlying mutations with different effects on LDL-C levels, and highlights the need for caution in interpreting historical LDL-C values. Furthermore, some patients with clinical FH (10%-40%) lack an identified disease-causing mutation.

A genetic diagnosis is highly desirable since the phenotype of severe hypercholesterolemia is highly overlapping.

Actually 4 genes have been described being involved in the disease. The most common genetic defects in FH are LDLR mutations (prevalence 1 in 500, depending on the population), ApoB mutations (prevalence 1 in 1000), PCSK9 mutations (less than 1 in 2500) and LDLRAP1. The related disease sitosterolemia, which has many similarities with FH and also features cholesterol accumulation in tissues, is due to ABCG5 and ABCG8 mutations.

LDL receptor The LDL receptor gene is located on the short arm of chromosome 19 (19p13.1-13.3). It comprises 18 exons and spans 45 kb, and the protein gene product contains 839 amino acids in mature form. A single abnormal copy (heterozygote) of FH causes cardiovascular disease by the age of 50 in about 40% of cases. Having two abnormal copies (homozygote) causes accelerated atherosclerosis in childhood, including its complications. The plasma LDL levels are inversely related to the activity of LDL receptor (LDLR). Homozygotes have LDLR activity of less than 2%, while heterozygotes have defective LDL pro-cessing with receptor activity being 2-25%, depending on the nature of the mutation. Over 1000 different mutations are known.

Apolipoprotein B Apolipoprotein B, in its ApoB100 form, is the main apolipoprotein, or protein part of the lipoprotein particle. Its gene is located on the second chromosome (2p24-p23) and is be-tween 21.08 and 21.12 Mb long. FH is often associated with the mutation of R3500Q, which causes replacement of arginine by glutamine at position 3500. The mutation is located on a part of the protein that normally binds with the LDL receptor, and binding is reduced as a result of the mutation. Like LDLR, the number of abnormal copies determines the severity of the hypercholesterolemia.

PCSK9 Mutations in the proprotein convertase subtilisin/kexin type 9 (PCSK9) gene were linked to autosomal dominant (i.e. requiring only one abnormal copy) FH in a 2003 report. The gene is located on the first chromosome (1p34.1-p32) and encodes a 666 amino acid protein that is expressed in the liver. It has been suggested that PCSK9 causes FH mainly by reducing the number of LDL receptors on liver cells.

LDLRAP1 Abnormalities in the ARH gene, also known as LDLRAP1, were first reported in a family in 1973. In contrast to the other causes, two abnormal copies of the gene are required for FH to develop (autosomal recessive). The mutations in the protein tend to cause the production of a shortened protein. Its real function is unclear, but it seems to play a role in the relation between the LDL receptor and clathrin-coated pits. People with autosomal recessive hypercholesterolemia tend to have more severe disease than LDLR-heterozygotes but less severe than LDLR-homozygotes.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures
* Patients of both genders older than 2 months
* The patient has a diagnosis of a homozygous familial Hypercholesterolemia or a high grade suspicion for a homozygous familial Hypercholesterolemia

High grade suspicion present, if one or more inclusion criteria are valid:

* Positive family anamnesis for a homozygous familial hypercholesterolemia
* Xanthomas
* Corneal arcus
* High levels of plasma cholesterol
* Manifestations of premature coronary heart disease

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related procedures.
* Patients of both gender younger than 2 months
* No diagnosis of a homozygous familial hypercholesterolemia or no valid criteria for profound suspicion of a homozygous familial hypercholesterolemia

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a Homozygous familial Hypercholesterolemia or high-grade suspicion for Homozygous familial Hypercholesterolemia
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Sequencing of the Homozygous Familial Hypercholesterolemia disease related genes | 4 weeks
  Next-Generation Sequencing (NGS) of the following genes: LDLR, APoB, PCSK9 and LDLRAP1 will be performed. The mutation will be confirmed by Sanger sequencing.

SECONDARY OUTCOMES:
The Homozygous familial Hypercholesterolemia specific biomarker candidates finding | 24 months
  The quantitative determination of small molecules (molecular weight 150-700 kD, given as ng/μl) within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (4):
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - NIRMAN Navi Mumbai Institute of Research In Mental And Neurological Handicap/Pediatric Geneticist, Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided